CLINICAL TRIAL: NCT01275404
Title: ACT-ED: Acceptance and Commitment Therapy for Erectile Dysfunction Adaptation of ACT for Compliance With an Erectile Rehabilitation Program
Brief Title: Therapy for Erectile Dysfunction Adaptation of ACT for Compliance With an Erectile Rehabilitation Program
Acronym: ACT-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Center for Marital and Sexual Health of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-204
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
Keywords: Erectile Dysfunction; focus group; Quality of Life; 10-204
MeSH Terms: conditions — Prostatic Neoplasms; Erectile Dysfunction

ARMS (2):
- (SMRP) + nurse practitioner information phone calls (Experimental): Part A will use focus groups to gain feedback and refine the intervention. Part B will consist of a randomized pilot study where 70 men will be randomly assigned to one of two conditions: Sexual Medicine Rehabilitation (SMRP) plus nurse practitioner information phone calls and monitoring (SMRP+I), or SMRP plus the novel psychological intervention of Acceptance and Commitment Therapy for ED (SMRP+ACT-ED).
  Interventions: Behavioral: Sexual Medicine Rehabilitation Program + nurse practitioner information phone calls
- SMRP+ACT-ED (Experimental): Part A will use focus groups to gain feedback and refine the intervention. Part B will consist of a randomized pilot study where 70 men will be randomly assigned to one of two conditions: Sexual Medicine Rehabilitation (SMRP) plus nurse practitioner information phone calls and monitoring (SMRP+I), or SMRP plus the novel psychological intervention of Acceptance and Commitment Therapy for ED (SMRP+ACT-ED).
  Interventions: Behavioral: Sexual Medicine Rehabilitation Program + Acceptance and Commitment Therapy for Erectile Dysfunction

INTERVENTIONS:
Behavioral: Sexual Medicine Rehabilitation Program + nurse practitioner information phone calls — Baseline Assessment which is 90-minute patient focus group interviews. SMRP, provided to all participating patients, consists of the following steps: 1) An introductory visit with SMRP Director, Dr. Mulhall, to orient the patient to post-surgery erectile rehabilitation and assess the patient"s success with PDE-5 inhibitors; 2) Penile injection training provided by a NP over two visits, with follow-up calls as necessary until injection method and dose are deemed correct; 3) Follow-up visits with Dr. Mulhall every 4 months to monitor progress with rehabilitation. Study assessments will be administered at baseline, at 4-8 months post baseline (follow up 1) and 4-8- months post follow up 1 (follow up 2).
  Arms: (SMRP) + nurse practitioner information phone calls
Behavioral: Sexual Medicine Rehabilitation Program + Acceptance and Commitment Therapy for Erectile Dysfunction — Baseline Assessment which is 90-minute patient focus group interviews. SMRP+ACT-ED will receive four individual ACT-ED counseling sessions (60 minutes each) over a period of approximately four months, and will also be followed up with questionnaires 4 and 8 months post baseline These sessions focus on the four core elements of ACT: values, acceptance, exposure, and commitment. Study assessments will be administered at baseline, at 4-8 months post baseline (follow up 1) and 4-8- months post follow up 1 (follow up 2).
  Arms: SMRP+ACT-ED

SUMMARY:
The investigators know that treatment for prostate cancer and erectile dysfunction can impact sexual health and quality of life. They want to learn how the treatment affects one's emotional and social well-being.

They have developed a new type of counseling. Cancer patients seek counseling for lots of reasons. It often helps them cope because they can express their feelings with a trained professional. They hope that this counseling will teach patients skills that they can use to comply with erectile treatment programs, improve their sexual health and quality of life. These skills may also improve physical and emotional well-being. As part of this study they will ask the patient to provide feedback on the proposed counseling.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Men who are 1 to 3 years post radical prostatectomy for early stage prostate cancer
* Participated in penile injection program
* Are able to speak, read, write and understand English well enough to complete study assessment and communicate with an English speaking therapist

Part B

* Men who are up to 9 months post radical prostatectomy.
* Had good erectile functioning pre-surgery (i.e., 24 or greater on the IIEF Erectile Function Domain (EFD) score), graded their erections as a 1 or 2 on the standard 5 point Urology Erectile Function scale) or have a score of 7 or greater on the 1-10 pre-surgery erectile function scale on the SMRP assessment)
* Seen at MSKCC"s Sexual Medicine Rehabilitation Program (SMRP)
* Advised by the clinical staff of the SMRP to start penile injections.

Exclusion Criteria:

Part A

* Recurrence or progression of disease,
* Specific injection phobia (self report)
* A history of bipolar disorder or psychotic disorder (determined from self-report and/or chart review)
* Current major depression (determined by self report and/or clinician observation and assessment) that would preclude from giving informed consent or being an active participant in a focus group

Part B

* Specific injection phobia (self report)
* A history of bipolar disorder or psychotic disorder (determined from self-report and/or chart review)
* Current major depression (determined by self report and/or clinician observation and assessment) that would preclude from giving informed consent or being an active participant in a therapeutic session.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-12-28 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
To investigate the feasibility | 2 years
  acceptability, tolerability and adherence) of adapted ACT psychotherapy treatment integrated into an erectile rehabilitation program (i.e., ACT-ED).

SECONDARY OUTCOMES:
To investigate the impact of ACT-ED | 2 years
  on penile injection compliance, ED treatment satisfaction, sexual functioning, sexual self-esteem, ED bother, depression symptoms, acceptance and self-awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm